CLINICAL TRIAL: NCT02277847
Title: A Phase IV, Randomized Study to Evaluate the Safety and Efficacy of Idarubicin at Different Dosages Combined With Cytarabine as Induction Therapy for Newly Diagnosed Acute Myeloid Leukaemia
Brief Title: Idarubicin at Different Dosages as Induction Therapy for Newly Diagnosed Acute Myeloid Leukaemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDREC.[2010]017
Record Dates: First submitted 2014-08-25; First posted 2014-10-29 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: Idarubicin; Cytosine arabinoside; Efficacy; Safety
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Idarubicin; Cytarabine; Safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IDA 8mg/M2 (Experimental): IDA 8mg/M2 per day, D1-3. iv injection in 10 minutes;Ara-C：100-200mg/M2 per day, D1-7. administration advice: at first, 25 mg/M2 of Ara-C is given by fast intravenous injection, then 100 mg/M2 of Ara-C is given by continuous iv drip for 24 hours for successive 7 days.
  Interventions: Drug: Idarubicin(8mg/m2) and cytosine arabinoside
- IDA 10mg/M2 (Active Comparator): IDA 10mg/M2 per day, D1-3. iv. injection in 10mimutes;Ara-C：100-200mg/M2 per day, D1-7. administration advice: at first, 25 mg/M2 of Ara-C is given by fast intravenous injection, then 100 mg/M2 of Ara-C is given by continuous iv drip for 24 hours for successive 7 days.
  Interventions: Drug: Idarubicin(10mg/m2), cytosine arabinoside

INTERVENTIONS:
Drug: Idarubicin(8mg/m2) and cytosine arabinoside — IDA 8mg/M2 per day, D1-3. iv injection in 10 minutes;Ara-C：100-200mg/M2 per day, D1-7. administration advice: at first, 25 mg/M2 of Ara-C is given by fast intravenous injection, then 100 mg/M2 of Ara-C is given by continuous iv drip for 24 hours for successive 7 days.
  Other Names: Idarubicin; Cytosine arabinoside; Acute myeloid leukemia; Safety; Efficacy
  Arms: IDA 8mg/M2
Drug: Idarubicin(10mg/m2), cytosine arabinoside — IDA 10mg/M2 per day, D1-3. iv. injection in 10mimutes;Ara-C：100-200mg/M2 per day, D1-7. administration advice: at first, 25 mg/M2 of Ara-C is given by fast intravenous injection, then 100 mg/M2 of Ara-C is given by continuous iv drip for 24 hours for successive 7 days.
  Other Names: Idarubicin; Cytosine arabinoside; Acute myeloid leukemia; Safety; Efficacy
  Arms: IDA 10mg/M2

SUMMARY:
Study Design: Treatment, Randomized, Open Label, Parallel Assignment This study is an open randomized and controlled trial aiming at assessing the efficacy and safety of Idarubicin (IDA) at different doses of 8mg/m2 and 10mg/m2 combined with cytarabine as induction therapy for newly diagnosed Acute Myeloid Leukaemia (AML). All the recruited patients are allocated to group A ( 8mg/m2 group) or group B ( 10mg/m2) in random. It is advised that induction therapy should begain not late than 3 days after randomization. The regimens in detail can be refered in the therapy protocol.

DETAILED DESCRIPTION:
Idarubicin is a new generation of anthracyclines with high lipophilicity and is more permeable to cytomembrane and therefore is more cytotoxic to leukemic cells. It can pass through the blood brain barrier easily. so IDA has more advantages over other anthracyclines in prolonging the overall survival for AML. The induction therapy with idarubicin and cytarabine is now the first-line induction regimen for AML. Many clinical trails have indicated that the dosage of IDA is positively correlated with its effectiveness. But in China IDA has been used in varied dosages ranging from 6 to 12 mg/m2. In most Chinese hospitals, the usual dosage range of IDA is from 6 to 8 mg/m2 which may contribute to the much lower 5-year survival rates of AML reported in Chinese medical literature than those in foreign literature. What is the suitable dosage of IDA as induction therapy for Chinese AML population with the best efficacy but the lest increase of side effects? Till now there is no retrospective, randomized and multicentered clinical trails to answer this question on remission-inducing dosages of IDA. All the existing trials till now are just small- sampled , single-centered , retrospective and non-randomized which can not provide strong evidences .

This study aims at comparing two induction doses of 8mg/m2 and 10mg/m2 of IDA with the method of prospective randomized and multi-centered trial.The two doses of IDA have been used in many Chinese hospitals for many years, its effectiveness and safety have been recognized. This trail aims at the and side effects of IDA during induction therapy and its effect on the long-term survival of Chinese AML population, so it can provide strong evidences for optimal dosage of IDA for Chinese AML population.It can not only reduce the waste of medical social resources but also produce good social and economic benefits.

ELIGIBILITY:
Inclusion Criteria:

* Age: 14~60 years old;no gender limit.
* Diagnosis: according to the diagnosis standards of AML( with the exception of M3 ) ( according to 2008 WHO diagnosis criteria of AML ).
* Performance status is not bad with Eastern Cooperative Oncology Group (ECOG) score ≤3.
* Research subjects must sign the informed consent documents.

Exclusion Criteria:

* Chronic myelogenous leukemia (CML) in crisis phase.
* AML transformed from other myeloproliferative diseases.
* Be accompanied with other progressing neoplasms.
* With severe malfunction of liver, lungs, kidneys or heart: the plasma levels of direct bilirubin, indirect bilirubin, alanine transaminase, aspartate transaminase and serum creatinine all are 2 times higher than normal, cardiac function is above grade II.
* With severe infection.

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Estimated)
Dates: Start 2010-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Overall survival(OS) and Disease free survival rate (DFS) | Within 5 years after randomization

SECONDARY OUTCOMES:
Induction remission rate | Within one month after induction therapy

OTHER OUTCOMES:
safety assessment (infection rate during induction therapy, liver and kidney toxicity, therapy related mortality, recovery time of blood count) | Randomization until death or two years post last subject last treatment visit (or clinical cutoff)

CONTACTS AND LOCATIONS:
Overall Officials: Xin Du, MD.PhD, Principal Investigator — Guangdong Provincial People's Hospital

REFERENCES:
- [Result] Yamashita T, Fukushima T, Ueda T. Pharmacokinetic self-potentiation of idarubicin by induction of anthracycline carbonyl reducing enzymes. Leuk Lymphoma. 2008 Apr;49(4):809-14. doi: 10.1080/10428190801947526. PMID 18398750
- [Result] Tsimberidou A, Estey E, Cortes J, Thomas D, Faderl S, Verstovsek S, Garcia-Manero G, Keating M, Albitar M, O'Brien S, Kantarjian H, Giles F. Gemtuzumab, fludarabine, cytarabine, and cyclosporine in patients with newly diagnosed acute myelogenous leukemia or high-risk myelodysplastic syndromes. Cancer. 2003 Mar 15;97(6):1481-7. doi: 10.1002/cncr.11239. PMID 12627513
- [Result] Russo D, Malagola M, de Vivo A, Fiacchini M, Martinelli G, Piccaluga PP, Damiani D, Candoni A, Michielutti A, Castelli M, Testoni N, Ottaviani E, Rondoni M, Pricolo G, Mazza P, Zuffa E, Zaccaria A, Raspadori D, Bocchia M, Lauria F, Bonini A, Avanzini P, Gugliotta L, Visani G, Fanin R, Baccarani M. Multicentre phase III trial on fludarabine, cytarabine (Ara-C), and idarubicin versus idarubicin, Ara-C and etoposide for induction treatment of younger, newly diagnosed acute myeloid leukaemia patients. Br J Haematol. 2005 Oct;131(2):172-9. doi: 10.1111/j.1365-2141.2005.05745.x. PMID 16197446
- [Result] Chaleff S, Hurwitz CA, Chang M, Dahl G, Alonzo TA, Weinstein H. Phase II study of 2-chlorodeoxyadenosine plus idarubicin for children with acute myeloid leukaemia in first relapse: a paediatric oncology group study. Br J Haematol. 2012 Mar;156(5):649-55. doi: 10.1111/j.1365-2141.2011.08976.x. PMID 22512017
- [Result] Telek B, Rejto L, Kiss A, Batar P, Remenyi G, Szasz R, Ujj ZA, Udvardy M. [Current treatment of acute myeloid leukaemia in adults]. Orv Hetil. 2012 Feb 19;153(7):243-9. doi: 10.1556/OH.2012.29304. Hungarian. PMID 22318524